CLINICAL TRIAL: NCT00466310
Title: Metabolic Signatures and Biomarkers in First Episode and Recurrent Patients With Schizophrenia in Comparison to Healthy Controls
Brief Title: Metabolic Signatures and Biomarkers in Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00008577; 8370 (Other: Duke legacy protocol number)
Record Dates: First submitted 2007-04-25; First posted 2007-04-27 (Estimated); Results first posted 2013-01-03 (Estimated); Last update posted 2014-07-25 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Metabolomics
MeSH Terms: conditions — Schizophrenia | interventions — Aripiprazole; Risperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Aripiprazole for 4 weeks (Active Comparator): Blood is drawn for baseline. 20 Subjects are randomly assigned to receive Aripiprazole for weeks weeks with a starting dose of 10mg/day and the dose will be titrated to a maximum of 30mg /day based on effectiveness and tolerability. After 4 weeks of treatment, blood will be drawn again for metabolomics.
  Interventions: Drug: Aripiprazole
- Risperidone for 4 weeks (Active Comparator): Blood will be drawn for baseline evaluation. 20 Subjects will be randomly assigned to receive risperidone at a starting dose of 2mg/day, and can be increased to 6mg/day based on response of the subject. After 4 weeks of medication, blood is drawn again.
  Interventions: Drug: Risperidone
- Healthy volunteers (Other): Fasting blood samples will be drawn from healthy volunteers to match age, race and gender with the research subjects for comparison.
  Interventions: Other: Healthy volunteers

INTERVENTIONS:
Drug: Aripiprazole — Aripiprazole for 4 weeks
  Other Names: Abilify
  Arms: Aripiprazole for 4 weeks
Drug: Risperidone — Subjects will be randomized to risperidone for 4 weeks
  Other Names: Risperdal
  Arms: Risperidone for 4 weeks
Other: Healthy volunteers — Healthy volunteers
  Arms: Healthy volunteers

SUMMARY:
We plan to use a metabolomics lipid platform to map biochemical signatures in unmedicated schizophrenic patients prior to and 4 weeks post treatment with the antipsychotic drug aripiprazole and compare that to lipid perturbations induced by risperidone. These drugs have inherently different risk for metabolic adverse effects and patients respond to them differently. Metabolic signatures for the drugs capture significant biochemical information that could explain part of the basis for varied drug response within individuals and will highlight pathways implicated in drug action and in disease pathogenesis possibly enabling new drug design strategies. In addition, we will compare patients to healthy controls at baseline in regard lipid profiles.

DETAILED DESCRIPTION:
Schizophrenia (SCH) is a devastating mental disease that affects the human population worldwide with an incidence of about 1%. Most individuals with this illness benefit from long-term pharmacotherapy, however, the therapeutic effects of antipsychotic treatment are inconsistent, incomplete, and often countered by significant side-effects associated with long-term physical morbidity (e.g., tardive dyskinesia, obesity, hyperglycemia, hyperlipidemia. Metabolomics is a powerful new technology that provides a snap shot of biochemical pathways at a particular point in time. It has been earmarked as an important area to develop under the NIH roadmap initiative. We plan to use this platform to map biochemical signatures in unmedicated schizophrenic patients prior to and 4 weeks post treatment with the antipsychotic drug aripiprazole and compare that to lipid perturbations induced by risperidone. These drugs have inherently different risk for metabolic adverse effects and patients respond to them differently. Metabolic signatures for the drugs capture significant biochemical information that could explain part of the basis for varied drug response within individuals and will highlight pathways implicated in drug action and in disease pathogenesis possibly enabling new drug design strategies.In addition, we will compare patients to healthy controls at baseline in regard lipid profiles, to assess whether lipid profiles differ between unmedicated schizophrenia patients and healthy controls.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Diagnosis of schizophrenia
* Actively psychotic
* No more than a single dose of antipsychotic in the preceding 2 weeks

Exclusion Criteria:

* Mental retardation, epilepsy or history of head trauma
* Substance use disorder that explains the majority of the psychopathology
* Pregnant or lactating females

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2007-02; Primary Completion 2009-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rima Kaddurah-Daouk, MD, Principal Investigator — Duke University
Locations (1):
- John Umstead Hospital, Butner, North Carolina, United States

REFERENCES:
- [Background] Storey JD, Tibshirani R. Statistical significance for genomewide studies. Proc Natl Acad Sci U S A. 2003 Aug 5;100(16):9440-5. doi: 10.1073/pnas.1530509100. Epub 2003 Jul 25. PMID 12883005
- [Result] Kaddurah-Daouk R, McEvoy J, Baillie R, Zhu H, K Yao J, Nimgaonkar VL, Buckley PF, Keshavan MS, Georgiades A, Nasrallah HA. Impaired plasmalogens in patients with schizophrenia. Psychiatry Res. 2012 Aug 15;198(3):347-52. doi: 10.1016/j.psychres.2012.02.019. Epub 2012 Apr 16. PMID 22513041

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Unmedicated patients treated for a first psychotic episode (n = 20), and patients treated for psychotic relapse of schizophrenia or schizoaffective disorder(n = 20).
  Controls who had no personal history of psychotic illness or relatives with psychotic illnesses,(n = 31). Individuals receiving treatment for diabetes or hyperlipidemia were excluded.
Groups:
- First Episode Schizophrenics: Schizophrenia subjects with no prior episodes
- Recurrent Episode Schizophrenics: Schizophrenia subjects with at least one prior episode
- Healthy Volunteers: Fasting blood samples were drawn at baseline from 31 healthy matched controls.
Period: Overall Study
Arm/Group | First Episode Schizophrenics | Recurrent Episode Schizophrenics | Healthy Volunteers
Started | 20 | 20 | 31
Completed | 20 | 20 | 31
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- First Episode Schizophrenics: These are subjects with no prior schizophrenic episodes
- Recurrent Episode Schizophrenics: These subjects have had at least one prior schizophrenic episode.
- Total: Total of all reporting groups
Arm/Group | First Episode Schizophrenics | Recurrent Episode Schizophrenics | Healthy Volunteers | Total
Number analyzed (Participants) | 20 | 20 | 31 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 31 | 71
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (9.8) | 36.6 (12.7) | 37.9 (9.1) | 33.63 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 25 | 37
  Male | 13 | 15 | 6 | 34
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 31 | 71

OUTCOME MEASURES:

1. Primary Outcome: Total Plasmalogen Levels in the Lipid Profile
Description: Plasmalogens are a subclass of glycerophospholipids and ubiquitous constituents of cellular membranes and serum lipoproteins. Several neurological disorders show decreased level of plasmalogens.
Time Frame: Baseline
Population: 17 of the 31 available controls were age and BMI matched to the schizophrenia subjects.
Measure: Mean (Standard Deviation); unit: nmoles/gram
Arm/Group | First Episode Schizophrenics | Recurrent Episode Schizophrenics | Healthy Volunteers
Number analyzed (Participants) | 20 | 20 | 17
nmoles/gram | 57.65 (14.37) | 59.57 (15.87) | 75 (19.17)
Statistical Analysis 1: Comparison: First Episode Schizophrenics vs Recurrent Episode Schizophrenics vs Healthy Volunteers; A wilcoxon rank sum test was performed comparing baseline plasmalogen values, comparing schizophrenia subjects vs controls.P values from this analysis were adjusted for false discovery rates by the method of Storey and Tribshiani; Test type: Superiority or Other; p = 0.0149, Wilcoxon (Mann-Whitney) — Unadjusted p value is .0041

ADVERSE EVENTS:
Arm/Group | First Episode Schizophrenics | Recurrent Episode Schizophrenics | Healthy Volunteers
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/31
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20 | 0/31

LIMITATIONS AND CAVEATS:
Limited to patients admitted to Psychiatric facility

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes